CLINICAL TRIAL: NCT03440320
Title: Online Education and Gentle Exercise Intervention
Acronym: MY-Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Arlene Schmid, Co-Prinicipal Investigator, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-7581H; R34AT009688 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-22 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Pain
Keywords: Caregiving Dyad; Pain-related Disability
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: Online intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Demographic data and measures will be collected by a blinded and trained research assistant.
  The assessor and participants will be blinded to the randomization. We will maintain assessor and participant blinding through established mechanisms (e.g., not discussing information or intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MY-Skills Intervention - online (Experimental): Participants will complete an 8-week, 16 session class. Each class will consist of approximately an hour of light exercise and an hour of education designed to meet the needs of a caregiving dyad with chronic pain.
  Interventions: Behavioral: MY-SKILLS - online
- MY-Plan control - online (Active Comparator): Participants will complete an 8-week, 16 session class. Each class will consist of approximately an hour of light exercise and an hour of education designed to meet the needs of a caregiving dyad with chronic pain.
  Interventions: Behavioral: MY-Plan control - online

INTERVENTIONS:
Behavioral: MY-SKILLS - online — Participants will complete an 8-week, 16 session class. Each class will consist of approximately an hour of yoga and an hour of self-management designed to meet the needs of a caregiving dyad with chronic pain
  Arms: MY-Skills Intervention - online
Behavioral: MY-Plan control - online — Participants will complete an 8-week, 16 session class. Each class will consist of approximately an hour of exercise and an hour of education designed to meet the needs of a caregiving dyad with chronic pain..
  Arms: MY-Plan control - online

SUMMARY:
Aim 1: Develop and manualize the Education and Gentle Exercise intervention. Using focus groups, clinical reasoning, literature, and findings from previously tested interventions of yoga and self-management, the researchers will develop, refine, and standardize the Education and Gentle Exercise intervention for chronic pain. In parallel, the researchers will develop a control group that includes exercise and health and wellness education. The expected outcomes include Education and Gentle Exercise intervention workbooks for participants and training and teaching manuals for interventionists leading the Education and Gentle Exercise intervention group and control group.

Aim 2: Assess feasibility and acceptability of an online intervention, the Education and Gentle Exercise and research procedures including planned assessments. In this small RCT, the researchers will examine feasibility and acceptability of the 8-week Education and Gentle Exercise procedures and intervention compared to an exercise and health and wellness education control group. Participants will include 30 caregiving dyads randomly assigned to the two groups (15 dyads for Education and Gentle Exercise, and 15 dyads for control group; N = 30 dyads/60 participants). The primary hypothesis is that Education and Gentle Exercise will be feasible and acceptable to caregiving dyads, as measured by benchmarks for recruitment, screening, attendance, and completion of assessments and intervention. Surveys will be administered and focus groups will be conducted to understand participant satisfaction and experiences with Education and Gentle Exercise. After each intervention session, interventionists, caregivers, and care recipients will rate their satisfaction with the session content and activities.

DETAILED DESCRIPTION:
The long-term goal of this study is to advance best practices in complementary and integrative health (CIH) to improve health for caregivers and individuals with chronic disabilities. This proposal is focused on merging exercise and education to improve pain for individuals in a caregiving dyad. The objective of this study is to develop and test the online Education and Gentle Exercise intervention, thus, addressing the critical need for innovative pain interventions focusing on the caregiving dyad. To achieve this objective and support a future randomized controlled trial (RCT), the researchers will conduct a mixed-methods study, including a small RCT.

Aim 1: Develop and manualize the Education and Gentle Exercise intervention. Using focus groups, clinical reasoning, literature, and findings from previously tested interventions of yoga and self-management, the researchers will develop, refine, and standardize the Education and Gentle Exercise intervention for chronic pain. In parallel, the researchers will develop a control group that includes exercise and health and wellness education. The expected outcomes include Education and Gentle Exercise intervention workbooks for participants and training and teaching manuals for interventionists leading the Education and Gentle Exercise intervention group and control group.

Aim 2: Assess feasibility and acceptability of online Education and Gentle Exercise and research procedures including planned assessments. In this small RCT, the researchers will examine feasibility and acceptability of the 8-week Education and Gentle Exercise procedures and intervention compared to an exercise and health and wellness education control group. Participants will be assigned to one of the the two groups. The primary hypothesis is that the online Education and Gentle Exercise intervention will be feasible and acceptable to caregiving dyads, as measured by benchmarks for recruitment, screening, attendance, and completion of assessments and intervention. Surveys will be administered and focus groups will be conducted online to understand participant satisfaction and experiences with Education and Gentle Exercise. After each intervention session, interventionists, caregivers, and care recipients will rate their satisfaction with the session content and activities. To assess change on the primary outcome (pain-related disability) and secondary outcome measures, members of the caregiving dyad will complete pre and post-assessments guided by the Biopsychosocial model.

ELIGIBILITY:
Inclusion Criteria:

Both members of the caregiving dyad:

* Chronic musculoskeletal pain, present for a minimum of three months
* Moderate or high levels of daily pain-related disability (BPI ≥ 5)
* Part of caregiving dyad
* Adults age 18 and over and able to speak English
* Score >4 out of 6 on the short Mini Mental Status Exam
* Ability to stand with or without an assistive device
* Sedentary lifestyle (i.e., any waking behavior characterized by an energy expenditure ≤1.5 metabolic equivalents while in a sitting or reclining posture)

Inclusion for care recipient only:

-Living at home in the community (with or without caregiver)

Inclusion for caregiver only:

* Identified as the primary caregiver
* Caregiver at least the past six months

Exclusion Criteria:

* Significant cardiovascular disease: New York Heart Association functional class 3 or 4 congestive heart failure; systolic blood pressure ≥ 180 or diastolic blood pressure ≥ 105 mmHg; myocardial infarction within 3 months, chest pain or dizziness with exercise
* Stroke, or Transient Ischemic Attack within 6 months
* Respiratory conditions requiring use of oxygen at home (i.e., COPD)
* Receiving or planning to receive, cancer treatment in the next 6 months
* Alzheimer's disease, dementia; expectation of death in the next 12 months
* In current physical rehabilitation, drug/alcohol treatment, or exercise research study
* Completed self-management education in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Schmid, PhD, Principal Investigator — Colorado State University; Christine Fruhauf, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmid AA, Fruhauf CA, Fox AL, Sharp JL, Portz JD, Leach HJ, Van Puymbroeck M. A pilot study to establish feasibility and acceptability of a yoga and self-management education intervention to support caregivers and care receivers with persistent pain. Front Rehabil Sci. 2024 Oct 3;5:1397220. doi: 10.3389/fresc.2024.1397220. eCollection 2024. PMID 39421567
- [Derived] Portz JD, Schmid A, Fruhauf C, Fox A, Van Puymbroeck M, Sharp J, Leach H. Acceptability of Online Yoga Among Individuals With Chronic Conditions and Their Caregivers: Qualitative Study. JMIR Form Res. 2023 May 24;7:e39158. doi: 10.2196/39158. PMID 37223971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MY-Skills Intervention - Online | MY-Plan Control - Online
Started | 18 | 14
Completed | 18 | 13
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Online Pilot, MY-Skills (Intervention), Caregivers: Participants in the MY-Skills program who provide the most care to their partner (other member of the dyad).
- Online Pilot, MY-Skills (Intervention), Care Receivers: Participants in the MY-Skills program who receive the most care from their partner (other member of the dyad).
- Online Pilot, MY-PLAN (Control), Caregivers: Participants in the MY-PLAN control group who provide the most care to their partner (other member of the dyad).
- Online Pilot, MY-PLAN (Control), Care Receivers: Participants in the MY-PLAN control group who receive the most care from their partner (other member of the dyad).
- Total: Total of all reporting groups
Arm/Group | Online Pilot, MY-Skills (Intervention), Caregivers | Online Pilot, MY-Skills (Intervention), Care Receivers | Online Pilot, MY-PLAN (Control), Caregivers | Online Pilot, MY-PLAN (Control), Care Receivers | Total
Number analyzed (Participants) | 9 | 9 | 7 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.33 (20.72) | 65.00 (18.97) | 37.57 (12.73) | 39.86 (21.04) | 52.19 (21.68)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: unreported data from one participant
  Participants
    number analyzed (Participants) | 9 | 9 | 7 | 6 | 31
    Female | 6 | 8 | 1 | 6 | 21
    Male | 3 | 1 | 6 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 7 | 7 | 4 | 5 | 23
  Unknown or Not Reported | 1 | 1 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 7 | 8 | 6 | 7 | 28
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
PROMIS-29 Profile v2 [Mean (Standard Deviation); unit: units on a scale] — Population: unreported data from one participant
  units on a scale
    number analyzed (Participants) | 9 | 9 | 6 | 7 | 31
    (all) | 78.56 (12.05) | 80.22 (16.08) | 69.17 (12.47) | 88.57 (3.95) | 79.48 (13.33)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory
Description: Change from baseline in pain on the Brief Pain Inventory scale following the 8-week intervention. The measure scores range from 0 to 10 with higher scores indicating more severe pain and greater interference. Reported scores indicate the change in scores from baseline to 8-weeks (after the intervention), with a potential range from -10 to 10. Negative scores would indicate and improvement (decrease) in pain severity and interference, while positive scores indicate an increase in pain severity and interference.
  Caregiver and care receiver completed the assessment on their own pain.
Time Frame: Administered at baseline and again following the 8-week intervention
Measure: Mean (Standard Deviation); unit: Change in score of units on a scale
Arm/Group | Online Pilot, MY-Skills (Intervention), Caregivers | Online Pilot, MY-Skills (Intervention), Care Receivers | Online Pilot, MY-PLAN (Control), Caregivers | Online Pilot, MY-PLAN (Control), Care Receivers
Number analyzed (Participants) | 9 | 8 | 6 | 7
Change in score of units on a scale | 0.23 (1.34) | -0.29 (1.63) | -1.38 (1.83) | -1.32 (1.87)

ADVERSE EVENTS:
Time Frame: 9 months, the span of time we conducted every intervention cohort
Description: Serious adverse event information collected and evaluated by our Institutional Review Board.
Arm/Group | MY-Skills Intervention - Online | MY-Plan Control - Online
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/14
Other Adverse Events (participants affected / at risk) | 0/18 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MY-Skills Intervention - Online (N=18) | MY-Plan Control - Online (N=14)
Extreme leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — SAE did not happen during active intervention/control. Participant hospitalized for extreme leg pain, received care, and released. Returned the next week, resumed sessions with med clearance. The SAE was deemed not related to the study by the IRB.
High blood pressure (Cardiac disorders) | 1 (1) | 0 (0) — SAE did not occur during active intervention/control. Participant hospitalized for high blood pressure and dizziness, received care and released with new medication. Resumed sessions with med clearance. SAE deemed not related to study by IRB.

LIMITATIONS AND CAVEATS:
Very specific inclusion and exclusion criteria (requiring high levels of pain severity and interference and low levels of physical activity) may have limited our ability to recruit a larger number of eligible individuals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03440320/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03440320/SAP_001.pdf
  • Informed Consent Form (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT03440320/ICF_002.pdf